CLINICAL TRIAL: NCT06051110
Title: Individual Patient Data Meta-analysis on Prehospital Risk Assessment in Patients Suspected of Non-ST-segment Elevation Acute Coronary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Pieter-Jan Vlaar, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: nWMO-2023.086
Record Dates: First submitted 2023-09-04; First posted 2023-09-22 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome; Non ST Segment Elevation Acute Coronary Syndrome
Keywords: EMS; POC-troponin; Combined risk scores; Prehospital
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Other): Patients who receive usual care by EMS protocols
  Interventions: Other: Usual care
- point-of-care troponin (Other): Patients in who risk-stratification was performed by the use of a point-of-care troponin in the EMS setting
  Interventions: Device: point-of-care troponin
- Combined risk scores (Other): Patients in who risk-stratification was performed by the use of a combined risk score in the EMS setting
  Interventions: Device: Combined risk score

INTERVENTIONS:
Device: Combined risk score — Prehospital risk stratification by the use of a combined clinical risk score including POC-troponin
  Arms: Combined risk scores
Other: Usual care — Prehospital risk stratification by EMS protocols
  Arms: Usual care
Device: point-of-care troponin — Prehospital risk stratification by the use of a POC-troponin
  Arms: point-of-care troponin

SUMMARY:
Patients with a non-ST-segment elevation acute coronary syndrome (NSTE-ACS) are currently transported and admitted to the nearest emergency department (ED) for risk stratification, diagnostic workup, and treatment. Recently, several prospective studies have been performed on the diagnostic performance of point-of-care (POC)-troponin and combined risk scores (CRS) for pre-hospital risk assessment and triage of NSTE-ACS patients. Also the first intervention trials on triage decisions based on POC troponin and CRS have been performed. Initial results are indicating that prehospital triage based on these diagnostic tools is feasible and safe, although sample sizes were relatively small and underpowered to detect differences in major adverse cardiac events (MACE). The objective of this individual patient data meta-analysis is to determine the diagnostic performance of POC troponin and combined risk scores for prehospital risk assessment and triage in suspected NSTE-ACS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suspected for NSTE-ACS;
2. Prospective study
3. Original data
4. Presenting prehospital (EMS)
5. Prehospital risk assessment using at least POC-troponin, performed and analyzed by EMS.
6. Outcome data available on in-hospital ACS or MACE within 30 days.

Exclusion Criteria:

1. Enrolling only a specific subpopulation from the general ACS population
2. Studies with less than 100 patients
3. Studies enrolling only patients with STEMI.
4. Studies published before 1995 / the pre-troponin era
5. Studies performed by general practitioners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the diagnosis NSTE-ACS | During index hospitalization, up to 1 day in the ED
  Diagnosis of NSTE-ACS (NSTEMI or unstable AP) during index hospitalization (as assessed by the treating physician)
MACE | Within 30 days
  All cause death, myocardial infarction, revascularization

SECONDARY OUTCOMES:
MACE | 1 week
  All cause death, myocardial infarction, revascularization
All cause death | Within 30 days and 1 year follow-up
The number of participants undergoing invasive coronary angiography | During or after index hospitalisation, up to 30 days
The number of participants undergoing coronary revascularisation | During or after index hospitalisation, up to 30 days
  percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
Alternative diagnoses other than NSTE-ACS | during 30 day follow-up after inclusion
  If no NSTE-ACS is diagnosed, what is the alternative diagnosis (such as pulmonary embolism, aortic dissection, pneumothorax)
Safety endpoints concerning intracoronary angiography and/or PCI | during 30 day follow-up after intracoronary angiography and/or PCI
  Bleeding complications
Safety endpoints concerning intracoronary angiography and/or PCI | during 30 day follow-up after intracoronary angiography and/or PCI
  Contrast-induced nephropathy Possible or definite stent thrombosis Ischemic stroke Death
Safety endpoints concerning intracoronary angiography and/or PCI | during 30 day follow-up after intracoronary angiography and/or PCI
  Possible or definite stent thrombosis
Safety endpoints concerning intracoronary angiography and/or PCI | during 30 day follow-up after intracoronary angiography and/or PCI
  Ischemic stroke
Safety endpoints concerning intracoronary angiography and/or PCI | during 30 day follow-up after intracoronary angiography and/or PCI
  Death
Health care utilization | Within 30 days after inclusion
  Number of ambulance transfers
Health care utilization | Up to 30 days after inclusion
  Duration of hospitalisation (days)
Health care utilization | Within 30 days after inclusion
  Number of double invasive coronary angiography procedures
Total health care costs | At 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pieter-Jan Vlaar, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina hospital Eindhoven, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Demandt JPA, Zelis JM, Koks A, Smits GHJM, van der Harst P, Tonino PAL, Dekker LRC, van Het Veer M, Vlaar PJ. Prehospital risk assessment in patients suspected of non-ST-segment elevation acute coronary syndrome: a systematic review and meta-analysis. BMJ Open. 2022 Apr 5;12(4):e057305. doi: 10.1136/bmjopen-2021-057305. PMID 35383078
- [Background] Sagel D, Vlaar PJ, van Roosmalen R, Waardenburg I, Nieuwland W, Lettinga R, van Barneveld R, Jorna E, Kijlstra R, van Well C, Oomen A, Bartels L, Anthonio R, Hagens V, Hofma S, Gu Y, Drenth D, Addink R, van Asselt T, van der Meer P, Lipsic E, Juarez Orozco L, van der Harst P. Prehospital risk stratification in patients with chest pain. Emerg Med J. 2021 Nov;38(11):814-819. doi: 10.1136/emermed-2020-210212. Epub 2021 Aug 9. PMID 34373266
- [Background] Camaro C, Aarts GWA, Adang EMM, van Hout R, Brok G, Hoare A, Rodwell L, de Pooter F, de Wit W, Cramer GE, van Kimmenade RRJ, Damman P, Ouwendijk E, Rutten M, Zegers E, van Geuns RM, Gomes MER, van Royen N. Rule-out of non-ST-segment elevation acute coronary syndrome by a single, pre-hospital troponin measurement: a randomized trial. Eur Heart J. 2023 May 14;44(19):1705-1714. doi: 10.1093/eurheartj/ehad056. PMID 36755110
- [Background] Tolsma RT, Fokkert MJ, van Dongen DN, Badings EA, van der Sluis A, Slingerland RJ, van 't Riet E, Ottervanger JP, van 't Hof AWJ. Referral decisions based on a pre-hospital HEART score in suspected non-ST-elevation acute coronary syndrome: final results of the FamouS Triage study. Eur Heart J Acute Cardiovasc Care. 2022 Feb 8;11(2):160-169. doi: 10.1093/ehjacc/zuab109. PMID 34849660
- [Background] Demandt JPA, Koks A, Haest R, Heijmen E, Thijssen E, Otterspoor LC, van Veghel D, El Farissi M, Eerdekens R, Vervaat F, Pijls NHJ, Veer MVT, Tonino PAL, Dekker LRC, Vlaar PJ. Prehospital triage of patients with suspected non-ST-segment elevation acute coronary syndrome: Rationale and design of the TRIAGE-ACS study. Contemp Clin Trials. 2022 Aug;119:106854. doi: 10.1016/j.cct.2022.106854. Epub 2022 Jul 18. PMID 35863696